CLINICAL TRIAL: NCT03854513
Title: Impact of Residual Renal Function on Complications in Chronic Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Hassan Mohyeldein, Principal investigator, Assiut University
Other Study IDs: Impact of HD on Kidneys
Record Dates: First submitted 2019-02-14; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Hemodialysis Complication
MeSH Terms: interventions — Kidneys, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- -Group 1 (anuric): patients on maintenance hemodialysis after 6 months to 1 year or more and urinary output less than 100ml / day
  Interventions: Device: dialysis machine
- Group 2 (good UOP): patients on maintenance hemodialysis after 6 months to 1 year or more and urinary output 400ml / day or more
  Interventions: Device: dialysis machine

INTERVENTIONS:
Device: dialysis machine — A machine used in dialysis that filters a patient's blood to remove excess water and waste products when the kidneys are damaged

SUMMARY:
Our aim is to study the impact of residual renal function on hemodialysis patients mortality and morbidity .

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a progressive loss in renal function over a period of months or years. As kidney function declines, there is progressive deterioration in mineral homeostasis manifesting as disruption of serum and tissue concentrations of phosphorus and calcium (Ca), as well as changes in circulating levels of hormones such as parathyroid hormone (PTH). These mineral and endocrine functions are critically important in the regulation of both initial bone formation during growth (bone modeling) and bone structure and function during adulthood (bone remodeling) Residual renal function (RRF) plays an important role in maintaining fluid balance, phosphorus control, nutrition, and removal of middle molecular uremic toxins. Decline of RRF also contributes significantly to anemia, inflammation, and malnutrition in patients on dialysis.

Inflammation and activation of acute-phase responses are common in chronic kidney disease patients.

The causes of inflammation in HD patients are multifactorial. Inflammatory reaction may originate from several sources, including graft or fistula infections, bioincompatible dialysis membrane, dialysate, endotoxin exposure, back filtration, chronic infections, and malnutrition. High-sensitivity C-reactive protein (hsCRP) assay is useful for sensitive detection of the inflammatory state.

Residual renal function (RRF) in patients with end-stage renal disease (ESRD) receiving renal replacement therapy is defined as the ability of native kidneys to eliminate water and uremic toxins. In clinical practice, it is considered synonymous with such parameters as daily diuresis and/or glomerular filtration rate (GFR). The optimal method to measure RRF has not been established . RRF remains important even after beginning of dialysis. RRF contributes significantly to the overall health and well-being of patients on dialysis Residual Renal (RRF) plays an important role in maintaining fluid balance, phosphorus control, nutrition, and removal of middle molecular uremic toxins and shows inverse relationships with valvular calcification and cardiac hypertrophy in patients on dialysis.

Decline in RRF also contributes significantly to anemia, inflammation, and malnutrition in patients on dialysis . RRF may allow for a reduction in the duration of hemodialysis (HD) sessions and the need for dietary and fluid restrictions in both patients on peritoneal dialysis (PD) and patients on HD. More importantly, the loss of RRF is a powerful predictor of mortality. Much of RRF is lost during the first 18 months of HD, and appears to depend on the primary cause(s) of kidney failure as well as on other patient-related and treatment-related factors

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal failure patients on maintenance hemodialysis after at least six months.

Exclusion Criteria:

1. Obstructive uropathy.
2. Heart failure.
3. Chronic liver disease( decompensated liver cirrhosis and ascites).

Ages: 25 Years to 45 Years | Sex: Male
Age Groups: Adult
Study Population: any populatin
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-26 (Estimated); Primary Completion 2020-02-15 (Estimated); Study Completion 2020-04-20 (Estimated)

PRIMARY OUTCOMES:
determine complications of hemodialysis on patients with chronic kidney disease | baseline
  impact of residual renal function on hemodialysis patients mortality and morbidity and imprtance of high residual renal function on patients lifespan
  - residual renal function will assess by GFR which assess by MDRD and creatinine clearance methods

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A. Sobh, Study Director — Assuit Univeristy

REFERENCES:
- [Background] Hu SL, Joshi P, Kaplan M, Lefkovitz J, Poenariu A, Dworkin LD, Michaud DS. Rapid Change in Residual Renal Function Decline Is Associated with Lower Survival and Worse Residual Renal Function Preservation in Peritoneal Dialysis Patients. Perit Dial Int. 2017 Jul-Aug;37(4):477-481. doi: 10.3747/pdi.2016.00211. PMID 28676514
- [Background] Cho HY, Hyun HS, Kang HG, Ha IS, Cheong HI. Prevalence of 25(OH) vitamin D insufficiency and deficiency in pediatric patients on chronic dialysis. Perit Dial Int. 2013 Jul-Aug;33(4):398-404. doi: 10.3747/pdi.2011.00246. Epub 2012 Dec 3. PMID 23209039
- [Background] Maksic D, Colic M, Stankovic-Popovic V, Radojevic M, Bokonjic D. Systemic and intraperitoneal proinflammatory cytokines profiles in patients on chronic peritoneal dialysis. Med Pregl. 2007;60 Suppl 2:53-7. PMID 18928158
- [Background] Kazmi WH, Gilbertson DT, Obrador GT, Guo H, Pereira BJ, Collins AJ, Kausz AT. Effect of comorbidity on the increased mortality associated with early initiation of dialysis. Am J Kidney Dis. 2005 Nov;46(5):887-96. doi: 10.1053/j.ajkd.2005.08.005. PMID 16253729